CLINICAL TRIAL: NCT04882839
Title: Open Label, Phase 2 Study for Evaluating the Feasibility, Safety and Efficacy of Psychotherapy Assisted Psilocybin for Treatment of Severe Obsessive Compulsive Disorder (OCD) in Drug and/or Psychotherapy Resistant Patients.
Brief Title: Evaluating the Feasibility, Safety and Efficacy of Psychotherapy Assisted Psilocybin for Treatment of Severe OCD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: MSICS PHARMA LTD (Unknown)
Responsible Party: Principal Investigator, ODED ARBEL, Principal Investigator and Head of Day Care Unit, Beersheva Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0003-20-MHC2; MOH_2025-02-20_009663 (Other: Isreali minestry of health (MOH))
Record Dates: First submitted 2021-04-08; First posted 2021-05-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-02

CONDITIONS: Obsessive-compulsive Disorder
Keywords: obsessive compulsive disorder; psilocybin
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active participants (Experimental): Participants undertaking to full therapeutic protocol including psychotherapy sessions and Psilocybin sessions
  Interventions: Combination Product: psychotherapy assisted psilocybin

INTERVENTIONS:
Combination Product: psychotherapy assisted psilocybin — psychotherapy for patients while under the influence of psilocybin

SUMMARY:
Obsessive-compulsive disorder (OCD) is a neuropsychiatric disorder characterized by recurrent distressing thoughts and substantial anxiety, accompanied by repetitive behaviors or mental rituals. Individuals with OCD often have diminished quality of life, and functional impairment . The disorder cause high personal, societal and economic costs . Current available treatments for OCD show moderate response rate and high rate of symptom relapse. The purpose of the current study is to explore new alternative options for the treatment of OCD that can widely and continuously benefit patients. Specifically, The aim of this study is to investigate the feasibility, safety and efficacy of psychotherapy assisted psilocybin for treatment of severe OCD. Previous research has shown safety of treatment and high efficacy in reduction of anxiety and depression symptoms. However, only one study has evaluated the use of psilocybin for OCD patients. The protocol includes 15 therapeutic sessions, of which 12 are one-hour sessions for psychological preparation and integration, and three are eight hours' experiential sessions under the influence of psilocybin. The research will include 15 participants diagnosed with severe OCD, with at least one treatment failure. Assessments will be based on comparing ratings of the main outcome measure (Y-BOCS), at baseline, at the middle and at end of treatment. Other assessments will include data on side effects- to evaluate safety, and possible spiritual variables underlying change in symptoms via standardized questionnaires.

DETAILED DESCRIPTION:
Background and research rationale:

Obsessive-compulsive disorder (OCD) is a neuropsychiatric disorder characterized by recurrent distressing thoughts and substantial anxiety, accompanied by repetitive behaviours or mental rituals performed to control or alleviate this anxiety. Individuals with OCD often have diminished quality of life, functional impairment , and cause substantial caregiver burden and personal and societal economic costs. Lifetime prevalence of OCD ranges between 1.9%-2.5%, with patients often not responding to the offered pharmacological or psychological treatment, and in extreme cases may even undergo neurosurgical interventions.

There are several possible physiological mechanisms leading to the development of OCD, which may indicate several possible effective treatment options. Nowadays there is a consensus that the dopaminergic and serotonergic pathways are central to the development of the disorder with the basal ganglia as the main area of its origin. Other brain areas involved in OCD are the orbitofrontal cortex and anterior cingulate cortex which are connected to the basal ganglia and are involved in regulating attention and awareness. Abnormal activity between these areas and other subcortical areas might explain why normally unconscious information processing, becomes consciousness, and requires additional resources for its regulation. It has also been suggested that the aversive emotional activity (anxiety, fear, disgust) experienced in OCD, relates to hyperactivity in the amygdala. The momentary relief brought on by the compulsive behaviour forms a positive feedback which perpetuate the disorder.

The gold standard of care for OCD today is a combination of selective serotonin reuptake inhibitors (SSRIs) and cognitive behavioural therapy (CBT). Most patients will experience at least some symptomatic relief with these interventions; however, relapse of symptoms occur in 40%-60% of patients and around 25% of patients are unresponsive to treatment . Other existing treatments (either pharmacological or neurosurgical) possess a higher risk for serious side effects. It is important to note that even for those patients who are responsive to treatment there are still significant residual, impairing symptoms. It thus seems that there is a real and immediate need to explore new alternative options for the treatment of OCD that can widely and continuously benefit patients, with lower risk and fewer side effects.

A new and promising prospect of treatment in mental health is the use of psychedelic substances, which interact with the serotonergic pathways and induce a powerful subjective experience with the potential for psychological transformation. Specifically, psilocybin has received attention in research as a promising alternative in the treatment of severe mental illness. Psilocybin is a prodrug which is quickly converted by the body to psilocin (4-OH-dimethyltryptamine), a 5-HT2A receptor partial agonist. Both psilocybin and psilocin, which have psychoactive properties, are naturally occurring in Psilocybe mushrooms and are structurally similar to the endogenous neurotransmitter serotonin.

As a direct 5-HT2A agonist, psilocybin has a unique therapeutic potential compared with other pharmacological treatment for OCD such as SSRIs. Animal studies have shown increased cognitive flexibility, associative learning, cortical plasticity, and anti-depressive effects in response to 5-HT2A activation.

The first current clinical research with psilocybin examined the safety and efficacy of psilocybin in the treatment of psychological distress in patients with terminal advanced-stage cancer. The double-blind, placebo-controlled research was conducted in the Los Angeles Biomedical Research Institute, Harbor-UCLA Medical Center (Torrance, California). Researchers concluded that psilocybin is safe and well tolerated at 0.2 mg/kg dose.

Following this research two different research groups, in Johns Hopkins University, and in New York University, have received FDA approval to administrate a higher dose of psilocybin in a similar clinical population. These trails have shown promising results for safety, psychological distress reduction, and significant improvement in anxiety and depression.

In their research, Griffiths and colleagues, examined the efficacy of psilocybin in reducing anxiety and depression in 51 patients suffering from a terminal end-stage cancer and experiencing symptoms of anxiety and depression. This randomized, double-blind, cross-over trial investigated the effects of a very low (placebo-like) dose (1 or 3 mg/70 kg) vs. a high dose (22 or 30 mg/70 kg) of psilocybin. No serious adverse events attributed to psilocybin administration occurred. There were transient moderate increases in systolic and/or diastolic blood pressure after psilocybin (in 34% of participants in the high-dose session and 17% of participants in the low-dose session), none of these episodes met criteria for medical intervention. Nausea or vomiting occurred in 15% of participants in the high-dose session. An episode of physical discomfort (any type) occurred in 21% of participants in the high-dose session and 8% in the low-dose session. Psychological discomfort (any type) occurred in 32% of participants in the high-dose session and 12% in the low-dose session. An episode of anxiety occurred in 26% of participants in the high-dose session and 15% in the low-dose session. One participant had a transient episode of paranoid ideation (2% of high-dose sessions). There were no cases of hallucinogen persisting perception disorder (HPPD) or prolonged psychosis. Across the two dose sequence groups, the overall rate of clinical response at 6 months was 78% and 83% for depression and anxiety, respectively, and the overall rate of symptom remission at 6 months for all participants was 65% and 57%, respectively.

Ross and colleagues conducted a double-blind, placebo-controlled, crossover trial, with 29 patients with cancer-related anxiety and depression that were randomly assigned and received treatment with single-dose psilocybin (0.3 mg/kg) or niacin (active placebo), both in conjunction with psychotherapy (before and after drug administration). The most common adverse effects were non-clinically significant elevations in blood pressure and heart rate (76%), headaches/migraines (28%), nausea (14%), transient anxiety (17%), and transient psychotic-like symptoms (7%). The medical and psychiatric adverse effects attributable to psilocybin are all known, were transient, and tolerable. There were no cases of prolonged psychosis or HPPD, and no participants required psychiatric hospitalization. Psilocybin produced immediate, substantial, and sustained improvements in anxiety and depression, this effect was sustained at 6.5 months follow-up.

These trails and others have shown safety of treatment and high efficacy in reduction of anxiety and depression symptoms with sustained effect at 6 months follow up. These findings taken together with the theoretical understanding of psilocybin mechanism of action and with the understanding of the neuro-psychological pathology of OCD, encourage investigating the potential of psilocybin as a novel significant treatment for this disorder. Research of beneficial effects of psilocybin for patients with OCD is in its infancy, but preliminary findings show potential efficacy in treatment of the disorder.

Matsushima and colleagues, used a mice model for OCD and found that psilocybin (both syntactic and in mushroom form), significantly inhibited compulsive behaviour (marble burying) without affecting locomotor activity. In addition, several case reports showed beneficial effects of psilocybin for people with OCD. For example, Leonard and Rapoport (1987) and Moreno and Delgado (1997) reported that among drug-users with OCD, there was a worsening of symptoms under the influence of cocaine, but a remission of symptoms for hours/ days following psilocybin use. Wilcox (2014) described a case in which a patient with OCD self-medicated with psilocybin, once every three weeks, experienced a preserved effect of reduced anxiety, obsessive thoughts, and compulsive behaviour. In another case report, a patient suffering from a body dysmorphic disorder (spending about 4 hours a day examining himself in the mirror), has experienced a significant reduction in distress and a notable change in body perception following multiple dosing of psilocybin.

Moreno et al. 2006 conducted a semi open-label trial examining the effect of psilocybin on nine participants with mild to severe OCD, which had at least one "treatment failure" defined as a lack of significant improvement after an adequate treatment. Doses were 25 (very low dose [VLD]), 100 (low dose [LD]), 200 (medium dose [MD]), and 300 (high dose [HD]) µg/kg. LD, MD, and HD were assigned in that order, and VLD was inserted randomly and in a double-blind fashion at any time after the first dose (LD). In measurements during the 24 hours after each dose all participants have experienced a significant relief in symptoms (23%-100% as measured by the Yale-Brown Obsessive-Compulsive Scale [YBOCS]) in at least one of the sessions. Two of the subjects reported that their symptomatic improvement lasted most of the following week after testing. One subject achieved long-term remission at the end of the 4 test sessions, as measured at 6-month follow-up. There was, however, no clear dose-response relationship to the change in YBOCS score and no correlation between YBOCS score reduction and the perceived intensity of the psychedelic experience.

These preliminary findings stress the need for further research to examine the efficacy of psilocybin in the treatment of OCD. In addition, the only clinical trial to date did not include psychotherapy for patients while under the influence of psilocybin. Earlier studies have shown that a preliminary therapeutic relationship before psilocybin administration increases the probability for a "peak experience" during sessions. Furthermore, two more recent studies have emphasized the importance of psychotherapy during and before psilocybin sessions, touching on 'intent' and formulating an early and strong therapeutic relationship. There is also a reference to the, "psychedelic afterglow", an effect lasting for days and even weeks after a psychedelic session during which there is a unique window for a meaningful transformative psychotherapeutic intervention, most likely owing to the increased psychological plasticity following a psychedelic experience.

The current study has two main goals: 1. Determine the safety and efficacy of psilocybin for patients suffering from OCD. 2. Elucidate the psychological mechanisms contributing to the beneficial effect of psilocybin on OCD symptoms.

Research Plan:

The current research aims to examine the feasibility, safety and efficacy of psychotherapy assisted psilocybin for treatment of severe OCD. The protocol includes 15 therapeutic sessions, of which 12 are one-hour sessions, and three are eight hours' experiential sessions (session 4,8,12) under the influence of psilocybin. In the first experiential session participants will receive a safety dose of 10mg/70kg. In the second and third sessions, participants will receive a therapeutic dose of 30mg/70kg. Three preparatory sessions will take place before the first experiential session, and three integration sessions will take place after each experiential session.

The research will include 15 participants, and will include the following phases:

Selection phase:

Research team will screen participants via phone interviews. Participants answering the inclusion criteria will be invited to receive and sign consent forms. Research member will collect demographics and health status data and register the participants according to study protocol.

Preparatory and final registration phase:

It is known that SSRIs have a counter effect on psilocybin; therefore, to allow a full effect of psilocybin it is necessary to avoid drug interaction and discontinue previous treatment. In a period of 4 weeks participants will undergo medication withdrawal under psychiatric supervision. During the 4 weeks period each participant will have 2-4 sessions (as needed) with the research psychiatrist, to supervise their clinical state. At the end of 4 weeks, a psychiatric evaluation will take place to determine readiness to begin psilocybin treatment.

Baseline assessment, and preparatory therapeutic sessions phase:

During the 5-6 weeks from registration, participants will have three preparatory psychotherapy sessions with a couple of therapists assigned to their treatment. Prior to their first psychotherapy session, participants will complete the first-baseline assessment of research questionnaires.

Treatment phase:

The treatment phase includes three experiential sessions with psilocybin (sessions 4, 8, 12), and three integration sessions after each experiential session. During this phase participants will complete three assessments using research questionnaires (sessions 2, 10, 15).

End of treatment and follow-up phase:

Primary outcome assessment will take place at the end of the last therapeutic session (no.15). Additional assessments will take place at three months, and six months/one-year follow-up.

Research procedure Participants will sign consent forms, before participating in the research treatment.

The treatment is based on 15 therapy sessions:

* Three preliminary sessions for establishing therapeutic alliance with the therapists and preparing the participant for the first experiential session.
* An 8-hour experiential session with a safety dose of psilocybin (10mg/70 kg). (V4)
* Participant will spend the night at the medical facility, under the supervision of a research member.
* A 1-hour session with the therapists, on the following morning (V5)
* Two integration sessions, and preparation for the next experiential session. (V6, V7)
* An 8-hour experiential session with a therapeutic dose of psilocybin (30mg/70 kg). (V8)
* Participant will spend the night at the medical facility, under the supervision of a research member.
* A 1-hour session with the therapists, on the following morning (V9)
* Two integration sessions, and preparation for the next experiential session. (V10, V11)
* An 8-hour experiential session with a therapeutic dose of psilocybin (30mg/70 kg). (V12)
* Participant will spend the night at the medical facility, under the supervision of a research member.
* A 1-hour session with the therapists, on the following morning (V13)
* Two integration and summary sessions. (V14, V15)

Possible discomfort:

It is possible that psilocybin and the experience it induces will cause some emotional or physical discomfort. Investigators will address all possible discomforts and appropriate measures to contain them, in the research safety instructions.

Research purpose:

The main objective of this research is to use standardized measuring tools to explore the safety and efficacy of psilocybin assisted psychotherapy in treating severe OCD symptoms. A secondary aim is to explore possible variables underlying change in symptoms.

Research objectives:

The main objective is to assess efficacy of psilocybin assisted psychotherapy in treating severe OCD symptoms. This assessment will be based on comparing ratings of the main outcome measure (Y-BOCS), at baseline (session 2) at the middle and at end of treatment (session 10, 15 respectively). A score under 14 or a reduction of 35% in the overall score will be considered as remission (Lewin, Nadai, Park, Goodman, Murphy & Stroch, 2011).

Secondary objectives: assessing safety by collecting data on side effects, and assessing possible spiritual variables underlying change in symptoms via standardized questionnaires and semi constructed interviews.

Safety:

The general safety goal is to assess occurrence and frequency of adverse events during treatment. This includes suicide ideation and/or behaviour, and adverse physiological or psychological responses. The safety of psilocybin use was previously proven in several clinical research.

Potential adverse effects:

In general, psychedelic drugs have low levels of physiological toxicity, and previous research indicate no evidence of toxicity, organ damage or neurophysiological disfunctions. Possible physiological effects experienced under the influence of psychedelic substances may include: dizziness, weakness, tremor, paresthesia, nausea, thirst, blurred vision, dilated pupils, and hyperreflexia. These somatic effects are dynamic and relatively minor, even when the psychological effect (sensory, perceptual, and cognitive) is strong/intense. The significant risk associated with psilocybin intake, is a subjective experience of fear and anxiety, panic, dysphoria and/or paranoia.

Recent clinical studies report a high safety level with no adverse effects. The high safety levels can be attributed to several control parameters described below, and to complying with safety guidelines in clinical psychotherapy with psychedelics. The use of psilocybin requires a significant psychotherapeutic holding of the subjective experience, that will provide a safe and supportive environment during the psychedelic experience. The safety guidelines in clinical psychotherapy with psychedelics describe the therapeutic presence and processes, as well as the set and settings needed to provide a supportive emotional and external environment.

Safety measures:

1. Controlling the quality of psilocybin and ensuring it is manufactured under GMP conditions.
2. Controlling for appropriate and adjusted dosage.
3. Controlling a strict protocol for screening eligible participants to the study (for details see inclusion-exclusion criteria section)
4. Recruiting professional and experienced psychotherapists with the appropriate training for clinical psychotherapy with psychedelics. Professionals will undergo a unique training to work with the psychotherapy protocol written for the current research.
5. Psychotherapists will work in pairs (a man and a woman), to provide an optimal holding space for each participant.
6. A proximity of a medical team for case of emergency.
7. Providing preparatory and integration sessions before and after the psilocybin sessions.
8. Preparing and using a comfortable and friendly room for the therapeutic session. The physical environment in which the treatment takes place should be suitable to the physical as well as the emotional safety of the participant. This means creating a lenient environment, which provides a pleasant and welcoming atmosphere, and may elicit a sense of intimacy and connection. As opposed to the environment of a hospital, a space like this supports and strengthens the participant's sense of safety and connectedness, thus helping him/her contain the intense psychedelic experience.
9. Guidelines for psychotherapy process: these guidelines are based on the humanistic perspective, and concern the characteristic of the therapeutic process:

   * A supportive, accepting, and non-judgmental presence of the therapist.
   * The importance of the therapeutic alliance and trust between participant and therapists.
   * A non-directive approach, supportive and gentle presence that stays with the participant's unfolding experience.
   * Viewing the mind as multi-dimensional, making space for the diverse dimensions of the internal experience: physical, emotional, and spiritual.
10. Maintaining a well-documented monitoring of the study and the participants status during the study period.
11. Monitoring physiological measure (blood pressure, heart rate and body temperature) during the psychedelic sessions with psilocybin: before taking the drug, an hour and a half after taking the drug, and 8 hours after. In case of anomalies physiological measures will be monitor more frequently.
12. Consulting and collaborating with other research teams with similar research interests, in NYU and Imperial College in London, UK.

ELIGIBILITY:
Inclusion Criteria:

* 1. DSM-5 diagnosis of OCD established by a trained clinician interview and confirmed by Mini International Neuropsychiatric Interview MINI (edition 7).

  2. Y-BOCS score of 16 or greater at evaluation 3. Treatment resistant- Patients; must have failed at least one medication and/or therapy trial of standard care treatment for OCD.

  4. Age: 18 Years to 65 Years 5. Has been off selective serotonin inhibitors for five half-lives of the drug plus 2 weeks.

  6. Must avoid starting new psychotherapy or psychiatric (medical) treatment during the study, without consulting the study team.

  7. Are willing to refrain from taking any psychiatric medications or recreational drugs during the study period.

  8. Must have a negative pregnancy test at study entry and prior to each experiential/ psychedelic session, if able to bear children, and must agree to use adequate birth control.

  9. Must be willing to sign a medical release form for the investigators to communicate directly with their therapist and doctors to confirm a medication and/or medical history. This is decided on a case by case basis upon the discretion of the PI.

  10. Must provide a contact (relative, spouse, close friend, or other caregiver) who is willing and able to be reached by the Clinical Investigators in the event of a participant becoming suicidal or any another relevant reason.

  11. Are willing to commit to medication dosing, experiential/ psychedelic sessions, psychotherapy and follow-up sessions and to complete the full evaluation.

Exclusion Criteria:

* 1. Personal or immediate family history of schizophrenia, bipolar affective disorder, delusion disorder, paranoid disorder, or schizoaffective disorder.

  2. Current (or last 12-month) substance abuse disorder. 3. Unstable neurological or medical condition. 4. Active suicidal intent or last 12-month suicidal attempt. 5. A history of violence, self-harm, or harm to another. 6. Any unstable medical condition that may render study procedures unsafe. 7. Positive urine pregnancy test at the time of screening. 8. Any use of psychedelic drugs within the prior 12 months. 9. Lack of ability to sign Informed consent. Exclusion Criteria during the study
  1. Any unusual reaction to any of the study procedures.
  2. A participant's request to stop his/ her participation in the study.
  3. Positive pregnancy test at any stage prior to the last psychedelic session

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS ) change from baseline | Baseline to 6-month follow-up
  severity of OCD symptoms- change from baseline
Obsessive-Compulsive Inventory-Revised (OCI-R) change from baseline | Baseline to 6-month follow-up
  OCD symptoms
Obsessional Beliefs Questionnaire (OBQ-20) change from baseline | Baseline to 6-month follow-up
  obsessive Beliefs
Beck Depression Inventory -II (BDI-II) change from baseline | Baseline to 6-month follow-up
  depression symptoms, will be measured by the Beck Depression Inventory
Beck Anxiety Inventory (BAI) change from baseline | Baseline to 6-month follow-up
  anxiety symptoms will be measured by the Beck Anxiety Inventory
Mini International Neuropsychiatric Interview (M.I.N.I.) change from baseline | Baseline to end of treatment
  psychopathological status will be measured by the Mini International Neuropsychiatric Interview

SECONDARY OUTCOMES:
5-Dimension - Altered States of Consciousness (5D-ASC) | 7 hours after drug administration
  Subjective altered states of consciousness will be measured by the 5-Dimension - Altered States of Consciousness
Mystical Experience Questionnaire (MEQ) | 7 hours after drug administration
  Changes in experiential aspects of psilocybin, will be measured by the Mystical Experience Questionnaire
Emotional Breakthrough Inventory (EBI) | Morning after drug administration
  Emotional breakthroughs will be measured by the Emotional Breakthrough Inventory
Persisting Effects Questionnaire (PEQ) | Baseline to 6-month follow-up
  Changes in spirituality, personal well-being, relationships, and emotions will be measured by the Persisting Effects Questionnaire
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | Baseline to 6-month follow-up
  Life satisfaction will be measured by the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form
Community Observer Questionnaire | Baseline to 6-month follow-up
  Changes in participants' behavior and attitudes will be measured by the structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Oded Arbel, MD, Principal Investigator — Beersheva Mental Health Center
Locations (1):
- Beer Sheva Mental Health Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No